CLINICAL TRIAL: NCT02555657
Title: A Randomized Open-Label Phase III Study of Single Agent Pembrolizumab Versus Single Agent Chemotherapy Per Physician's Choice for Metastatic Triple Negative Breast Cancer (mTNBC) - (KEYNOTE-119)
Brief Title: Study of Single Agent Pembrolizumab (MK-3475) Versus Single Agent Chemotherapy for Metastatic Triple Negative Breast Cancer (MK-3475-119/KEYNOTE-119)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-119; 2015-001020-27 (EudraCT Number); 153082 (Registry Identifier: JAPIC-CTI); MK-3475-119 (Other: Merck); KEYNOTE-119 (Other: Merck)
Record Dates: First submitted 2015-09-18; First posted 2015-09-21 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Triple Negative Breast Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Capecitabine; eribulin; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations (up to ~2 years). Qualified participants who receive first course of pembrolizumab but continue to experience disease progression may, at investigator's discretion, initiate a second course of pembrolizumab at 200 mg IV Q3W for up to 17 administrations (up to ~1 year).
  Interventions: Biological: pembrolizumab
- Chemotherapy (Active Comparator): Participants receive capecitabine, eribulin, gemcitabine, or vinorelbine as TPC in accordance with local regulations and guidelines.
  Interventions: Drug: capecitabine; Drug: eribulin; Drug: gemcitabine; Drug: vinorelbine

INTERVENTIONS:
Biological: pembrolizumab
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Drug: capecitabine
  Other Names: XELODA®
  Arms: Chemotherapy
Drug: eribulin
  Other Names: HALAVEN®
  Arms: Chemotherapy
Drug: gemcitabine
  Other Names: GEMZAR®
  Arms: Chemotherapy
Drug: vinorelbine
  Other Names: NAVELBINE®
  Arms: Chemotherapy

SUMMARY:
In this study, participants with metastatic triple negative breast cancer (mTNBC) will be randomly assigned to receive either single agent pembrolizumab or single agent chemotherapy chosen by the treating physician (Treatment of Physician's Choice, TPC) in accordance with local regulations and guidelines, consisting of either capecitabine, eribulin, gemcitabine, or vinorelbine. The primary study hypothesis is that pembrolizumab extends overall survival compared to TPC.

ELIGIBILITY:
Inclusion Criteria:

* Centrally confirmed Stage IV/M1 mTNBC
* Newly obtained tumor biopsy from metastatic site
* Central determination of programmed cell death ligand 1 (PD-L1) tumor status
* Received either one or two prior systemic treatments for metastatic breast cancer and have documented disease progression on or after the most recent therapy
* Previously treated with an anthracycline and/or taxane in the neoadjuvant/adjuvant or metastatic setting
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days prior to study start
* Adequate organ function

Exclusion Criteria:

* Participation in another clinical trial within 4 weeks
* Monoclonal antibody (mAb) for direct anti-neoplastic treatment within 4 weeks
* Chemotherapy, targeted small molecule therapy, or radiation therapy within at least 2 weeks
* Active autoimmune disease that required systemic treatment in the past 2 years
* Diagnosed with immunodeficiency or receiving systemic steroid therapy or another form of immunosuppressive therapy within 7 days
* Known additional malignancy that required treatment or progressed in last 5 years
* Known active brain metastases and/or carcinomatous meningitis
* Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-ligand-1 (anti-PD-L1), anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte associated protein 4 [CTLA-4], OX-40, CD137) or previously participated in any pembrolizumab (MK-3475) clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Cortes J, Lipatov O, Im SA, Goncalves A, Lee KS, Schmid P, Tamura K, Testa L, Ohtani S, Harbeck N, Loi S, Salgado R, Karantza V, Mejia J, Cristescu R, Loboda A, Nebozhyn M, Jelinic P, Huang L, Winer EP. Association of potential biomarkers with clinical outcomes in metastatic triple-negative breast cancer treated with pembrolizumab or chemotherapy. NPJ Breast Cancer. 2025 Oct 2;11(1):109. doi: 10.1038/s41523-025-00814-y. PMID 41038856
- [Derived] Essalihi A, Bouchra O, Khadiri K, Khadrouf Z, Karkouri M. Immunotherapy for triple-negative breast cancer: current trends and future prospects. J Egypt Natl Canc Inst. 2025 Jun 17;37(1):51. doi: 10.1186/s43046-025-00295-x. PMID 40526219
- [Derived] Schmid P, Lipatov O, Im SA, Goncalves A, Munoz-Couselo E, Lee KS, Tamura K, Testa L, Witzel I, Ohtani S, Turner N, Zambelli S, Harbeck N, Andre F, Dent R, Mejia JA, Zhou X, Haiderali A, Nguyen AM, Cortes J, Winer EP. Impact of pembrolizumab versus chemotherapy on health-related quality of life in patients with metastatic triple-negative breast cancer: results from the phase 3 randomised KEYNOTE-119 study. Eur J Cancer. 2023 Dec;195:113393. doi: 10.1016/j.ejca.2023.113393. Epub 2023 Oct 21. PMID 37976633
- [Derived] Winer EP, Lipatov O, Im SA, Goncalves A, Munoz-Couselo E, Lee KS, Schmid P, Tamura K, Testa L, Witzel I, Ohtani S, Turner N, Zambelli S, Harbeck N, Andre F, Dent R, Zhou X, Karantza V, Mejia J, Cortes J; KEYNOTE-119 investigators. Pembrolizumab versus investigator-choice chemotherapy for metastatic triple-negative breast cancer (KEYNOTE-119): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Apr;22(4):499-511. doi: 10.1016/S1470-2045(20)30754-3. Epub 2021 Mar 4. PMID 33676601
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response/progression or adverse events during the second pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures respectively.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations (up to ~2 years). Qualified participants who received first course of pembrolizumab but continued to experience disease progression may have, at investigator's discretion, initiated a second course of pembrolizumab at 200 mg IV Q3W for up to 17 administrations (up to ~1 year).
- Chemotherapy: Participants received capecitabine, eribulin, gemcitabine, or vinorelbine as single agent chemotherapy chosen by the treating physician (Treatment of Physician's Choice, TPC) in accordance with local regulations and guidelines.
Period: Overall Study
Arm/Group | Pembrolizumab | Chemotherapy
Started | 312 | 310
Treated | 309 | 292
Completed | 0 | 0
Not Completed | 312 | 310
Not completed — Death | 274 | 262
Not completed — Physician Decision | 0 | 1
Not completed — Sponsor Decision | 27 | 15
Not completed — Withdrawal by Subject | 11 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Chemotherapy | Total
Number analyzed (Participants) | 312 | 310 | 622
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (11.4) | 52.6 (11.2) | 52.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312 | 308 | 620
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 87 | 101 | 188
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 4 | 17
  White | 183 | 180 | 363
  More than one race | 12 | 12 | 24
  Unknown or Not Reported | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival in Participants With Programmed Cell Death Ligand 1 (PD-L1) With Combined Positive Score (CPS) ≥10
Description: Overall survival (OS) was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥10 who were included in a treatment group at randomization
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg IV every Q3W for up to 35 administrations (up to ~2 years).
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 96 | 98
Months | 12.7 [9.9 to 16.3] | 11.6 [8.3 to 13.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0574, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.57 to 1.06]

2. Primary Outcome: Overall Survival in Participants With PD-L1 CPS ≥1
Description: Overall survival (OS) was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥1 who were included in a treatment group at randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 203 | 202
Months | 10.7 [9.3 to 12.5] | 10.2 [7.9 to 12.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0728, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.69 to 1.06]

3. Primary Outcome: Overall Survival in All Participants
Description: Overall survival (OS) was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants who were included in a treatment group at randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 312 | 310
Months | 9.9 [8.3 to 11.4] | 10.8 [9.1 to 12.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.3802, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.82 to 1.15]

4. Secondary Outcome: Overall Response Rate Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With PD-L1 CPS ≥10
Description: Overall Response Rate (ORR), based on a Blinded Independent Central Review (BICR) assessment per RECIST 1.1, was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions).
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥10 who were included in a treatment group at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 96 | 98
Percentage of participants | 17.7 [10.7 to 26.8] | 9.2 [4.3 to 16.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0457, Miettinen & Nurminen method; Difference in percentages = 8.3, 95% CI 2-sided [-1.4 to 18.4]

5. Secondary Outcome: Overall Response Rate Per RECIST 1.1 in Participants With PD-L1 CPS ≥1
Description: Overall Response Rate (ORR), based on BICR assessment per RECIST 1.1, was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions).
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥1 who were included in a treatment group at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 203 | 202
Percentage of participants | 12.3 [8.1 to 17.6] | 9.4 [5.8 to 14.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.1752, Miettinen & Nurminen method; Difference in percentages = 2.9, 95% CI 2-sided [-3.3 to 9.2]

6. Secondary Outcome: Overall Response Rate Per RECIST 1.1 in All Participants
Description: as for outcome 5
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants who were included in a treatment group at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 312 | 310
Percentage of participants | 9.6 [6.6 to 13.4] | 10.6 [7.4 to 14.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.6629, Miettinen & Nurminen method; Difference in percentages = -1.0, 95% CI 2-sided [-5.9 to 3.8]

7. Secondary Outcome: Progression-Free Survival Per RECIST 1.1 in Participants With PD-L1 CPS ≥10
Description: Progression-Free Survival (PFS), based on BICR assessment per RECIST 1.1, was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥10 who were included in a treatment group at randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 96 | 98
Months | 2.1 [2.0 to 2.5] | 3.4 [2.3 to 4.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.7936, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.82 to 1.59]

8. Secondary Outcome: Progression-Free Survival Per RECIST 1.1 in Participants With PD-L1 CPS ≥1
Description: as for outcome 7
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥1 who were included in a treatment group at randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 203 | 202
Months | 2.1 [2.0 to 2.1] | 3.1 [2.3 to 4.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.9964, Regression, Cox; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.08 to 1.68]

9. Secondary Outcome: Progression-Free Survival Per RECIST 1.1 in All Participants
Description: as for outcome 7
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants who were included in a treatment group at randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 312 | 310
Months | 2.1 [2.0 to 2.1] | 3.3 [2.7 to 4.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 1.0000, Regression, Cox; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [1.33 to 1.92]

10. Secondary Outcome: Duration of Response Per RECIST 1.1 in Participants With PD-L1 CPS ≥10 Who Had a Confirmed Response
Description: For participants with PD-L1 CPS ≥10 who demonstrated a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, Duration of Response (DOR) was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on BICR.
Time Frame: Up to approximately 36 months (from time of first documented evidence of CR or PR through Final Analysis database cutoff date of 11-April-2019)
Population: All randomized participants with PD-L1 CPS ≥10, whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 17 | 9
Months | NA [2.2 to NA] — NA=Median DOR not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse | 7.1 [3.8 to NA] — NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse

11. Secondary Outcome: Duration of Response Per RECIST 1.1 in Participants With PD-L1 CPS ≥1 Who Had a Confirmed Response
Description: For participants with PD-L1 CPS ≥1 who demonstrated a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, Duration of Response (DOR) was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on BICR.
Time Frame: as for outcome 10
Population: All randomized participants with PD-L1 CPS ≥1, regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 25 | 19
Months | 12.2 [2.2 to NA] — NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse | NA [NA to NA] — NA=Median DOR not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR lower limit not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse

12. Secondary Outcome: Duration of Response Per RECIST 1.1 in All Participants Who Had a Confirmed Response
Description: For participants who demonstrated a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, Duration of Response (DOR) was defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions as well as an absolute increase of at least a 5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. DOR assessments were based on BICR.
Time Frame: as for outcome 10
Population: All randomized participants, regardless of whether or not they received study treatment, who demonstrated a confirmed response (CR or PR). Participants were included in the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 30 | 33
Months | 12.2 [2.2 to NA] — NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse | NA [NA to NA] — NA=Median DOR not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR lower limit not reached at time of data cutoff due to insufficient number of responding participants with relapse NA=DOR upper limit not reached at time of data cutoff due to insufficient number of responding participants with relapse

13. Secondary Outcome: Disease Control Rate Per RECIST 1.1 in Participants With PD-L1 CPS ≥10
Description: Disease Control Rate (DCR), based on BICR assessment per RECIST 1.1, was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) or Stable Disease for at least 24 weeks (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease [PD: At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD.])
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥10 who were included in a treatment group at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 96 | 98
Percentage of participants | 19.8 [12.4 to 29.2] | 17.3 [10.4 to 26.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.3388, Miettinen & Nurminen method; Difference in percentages = 2.3, 95% CI 2-sided [-8.7 to 13.5]

14. Secondary Outcome: Disease Control Rate Per RECIST 1.1 in Participants With PD-L1 CPS ≥1
Description: as for outcome 13
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants with PD-L1 CPS ≥1 who were included in a treatment group at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 203 | 202
Percentage of participants | 14.3 [9.8 to 19.9] | 15.8 [11.1 to 21.6]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.6701, Miettinen & Nurminen method; Difference in percentages = -1.6, 95% CI 2-sided [-8.6 to 5.5]

15. Secondary Outcome: Disease Control Rate Per RECIST 1.1 in All Participants
Description: as for outcome 13
Time Frame: Up to approximately 36 months (through Final Analysis database cutoff date of 11-April-2019)
Population: All participants who were included in a treatment group at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 312 | 310
Percentage of participants | 12.2 [8.8 to 16.3] | 18.7 [14.5 to 23.5]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.9877, Miettinen & Nurminen method; Difference in percentages = -6.5, 95% CI 2-sided [-12.2 to -0.8]

16. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to approximately 60 months
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 309 | 292
Participants | 285 | 281

17. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: as for outcome 16
Time Frame: Up to approximately 60 months
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 309 | 292
Participants | 14 | 16

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events (including first and second courses): Up to approximately 60 months
Description: All-cause mortality table includes all randomized participants. Serious and other AEs include participants who received at least 1 dose of study treatment. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug were excluded as AEs. Participants who received a second course of pembrolizumab per protocol were monitored for all-cause mortality and AEs separately.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg IV Q3W for up to 35 administrations (up to ~2 years).
- Chemotherapy: Participants received capecitabine, eribulin, gemcitabine, or vinorelbine as TPC in accordance with local regulations and guidelines.
- Pembrolizumab Second Course: Qualified participants who received the first course of pembrolizumab 200 mg IV Q3W for up to 35 administrations (up to ~2 years), but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q3W for up to 17 administrations (up to ~1 year).
Arm/Group | Pembrolizumab First Course | Chemotherapy | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 283/312 | 289/310 | 0/8
Serious Adverse Events (participants affected / at risk) | 65/309 | 60/292 | 1/8
Other Adverse Events (participants affected / at risk) | 259/309 | 263/292 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=309) | Chemotherapy (N=292) | Pembrolizumab Second Course (N=8)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (6) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (6) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Death (General disorders) | 0 (0) | 4 (4) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 8 (8) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation associated pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood corticotrophin abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Horner's syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=309) | Chemotherapy (N=292) | Pembrolizumab Second Course (N=8)
Anaemia (Blood and lymphatic system disorders) | 28 (31) | 46 (80) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 61 (146) | 0 (0)
Hypothyroidism (Endocrine disorders) | 25 (26) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 18 (18) | 15 (18) | 0 (0)
Constipation (Gastrointestinal disorders) | 50 (56) | 51 (59) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 29 (34) | 60 (83) | 1 (1)
Nausea (Gastrointestinal disorders) | 50 (63) | 89 (117) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (7) | 23 (24) | 0 (0)
Vomiting (Gastrointestinal disorders) | 23 (30) | 33 (44) | 0 (0)
Asthenia (General disorders) | 36 (40) | 38 (42) | 0 (0)
Fatigue (General disorders) | 55 (67) | 54 (61) | 1 (2)
Malaise (General disorders) | 9 (9) | 15 (17) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 22 (22) | 0 (0)
Oedema peripheral (General disorders) | 16 (17) | 14 (17) | 0 (0)
Pyrexia (General disorders) | 35 (46) | 34 (49) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (22) | 14 (20) | 0 (0)
Urinary tract infection (Infections and infestations) | 16 (18) | 20 (24) | 0 (0)
Alanine aminotransferase increased (Investigations) | 22 (25) | 24 (43) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 32 (39) | 28 (51) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (8) | 44 (144) | 0 (0)
Weight decreased (Investigations) | 10 (10) | 16 (16) | 0 (0)
White blood cell count decreased (Investigations) | 5 (11) | 30 (103) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 30 (31) | 38 (43) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (14) | 17 (21) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (46) | 24 (28) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (24) | 30 (33) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (20) | 24 (28) | 1 (1)
Dizziness (Nervous system disorders) | 14 (15) | 20 (21) | 0 (0)
Headache (Nervous system disorders) | 44 (61) | 34 (43) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 26 (28) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 19 (20) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (9) | 17 (18) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 53 (60) | 31 (33) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 (41) | 32 (39) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 43 (44) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 36 (47) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 35 (44) | 12 (12) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 23 (25) | 13 (14) | 0 (0)
Influenza like illness (General disorders) | 3 (4) | 4 (4) | 1 (3)
Blood bilirubin increased (Investigations) | 3 (3) | 8 (9) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (2):
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT02555657/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT02555657/SAP_002.pdf